CLINICAL TRIAL: NCT02426320
Title: Daily Interruption of Sedative Infusions in Mechanically Ventilated Children: A Randomized Pilot Study
Brief Title: Pilot Study for Sedation Interruption in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Davinia Withington (Other)
Responsible Party: Sponsor-Investigator, Davinia Withington, Pediatric Anesthesiologist and Intensivist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-011-PED
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Daily Sedative Interruption; Sedation Strategies; Sedation Protocols; Mechanical Ventilation; Sedation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sedation Interruption Protocol + standard sedation protocol (Active Comparator): Nurse directed protocols for administering sedation and/or analgesia, with daily interruption of sedation/analgesia
  Interventions: Other: Sedation Interruption Protocol
- Standard sedation protocol (Active Comparator): Nurse directed protocol for administering sedation and/or analgesia.
  Interventions: Other: Standard Sedation Protocol

INTERVENTIONS:
Other: Sedation Interruption Protocol
  Arms: Sedation Interruption Protocol + standard sedation protocol
Other: Standard Sedation Protocol
  Arms: Standard sedation protocol

SUMMARY:
The purpose of this study is to estimate the hypothesized benefit of sedation interruption protocol on mechanical ventilation duration and PICU length of stay. The study will evaluate recruitment rates, and adherence rates of such protocol.

DETAILED DESCRIPTION:
This is a prospective single-center, superiority, open randomized controlled trial comparing sedation interruption protocol and routine continuous sedation in mechanically ventilation (MV) children.

The study will be conducted in the twelve beds Pediatric Intensive Care Unit (PICU) at the Montreal Children's Hospital, a pediatric tertiary care and teaching hospital.

Patients will be enrolled prospectively within 24 hours of intubation and MV. After obtaining written consent patients will then be randomized to interrupted sedation or standard sedation protocol. The investigators will randomize using a computer-generated sequence of random numbers.

A Sedation protocol will be used for both groups to adjust continuous infusions of sedatives/analgesics to a targeted Comfort-Behavior scale. In the intervention group, sedation infusions will be interrupted daily at 8:00 AM, this interruption will be continued until the patient is under-sedated according to the Comfort Behavior scale goals or in the presence of symptoms of hemodynamic instability or respiratory distress. Then the patient will receive a bolus of sedation and the infusion will be restarted at a dose 50% less than the previous dose to return to the Comfort Score goal.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanically ventilated patients due to respiratory failure of multiple etiologies or after major surgical procedures for more than 24 hours.
* Sedation managed by benzodiazepines and opioids infusions

Exclusion Criteria:

* If sedation is required as part of medical management (Pulmonary hypertension, Increase intracranial pressure, Seizures
* Trauma & burn admissions
* Patients resuscitated from cardiac arrest
* Allergy to sedation (midazolam)
* Allergy to analgesia (fentanyl, morphine)
* Difficult airway including post-operative airway surgeries. (As deemed by ICU physician in charge)
* High frequency oscillator
* Special gas as inhaled nitric oxide, or isoflurane.
* Chronic ventilatory support
* Neuromuscular diseases
* Corrected Gestational age less than 37 weeks.
* Patients not expected to survive to discharge as per attending physician.
* Palliative care patients.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | At 30 days
  The number of eligible patients who provided informed consent to participate in the study divided by the total number of eligible patients who were asked for informed consent during the pilot study period over 1 year period.
Adherence Rate | At 30 days
Reasons for non-participation | At 30 days
Duration of mechanical ventilation in hours. | intraoperative
  Total number of hours between the moment patient was intubated to the moment of extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Conall Francoeur, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Christina Maratta, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Maryse Dagenais, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Schweickert WD, Gehlbach BK, Pohlman AS, Hall JB, Kress JP. Daily interruption of sedative infusions and complications of critical illness in mechanically ventilated patients. Crit Care Med. 2004 Jun;32(6):1272-6. doi: 10.1097/01.ccm.0000127263.54807.79. PMID 15187505
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Background] Anifantaki S, Prinianakis G, Vitsaksaki E, Katsouli V, Mari S, Symianakis A, Tassouli G, Tsaka E, Georgopoulos D. Daily interruption of sedative infusions in an adult medical-surgical intensive care unit: randomized controlled trial. J Adv Nurs. 2009 May;65(5):1054-60. doi: 10.1111/j.1365-2648.2009.04967.x. PMID 19399980
- [Background] Mehta S, Burry L, Cook D, Fergusson D, Steinberg M, Granton J, Herridge M, Ferguson N, Devlin J, Tanios M, Dodek P, Fowler R, Burns K, Jacka M, Olafson K, Skrobik Y, Hebert P, Sabri E, Meade M; SLEAP Investigators; Canadian Critical Care Trials Group. Daily sedation interruption in mechanically ventilated critically ill patients cared for with a sedation protocol: a randomized controlled trial. JAMA. 2012 Nov 21;308(19):1985-92. doi: 10.1001/jama.2012.13872. PMID 23180503
- [Background] Gupta K, Gupta VK, Jayashree M, Singhi S. Randomized controlled trial of interrupted versus continuous sedative infusions in ventilated children. Pediatr Crit Care Med. 2012 Mar;13(2):131-5. doi: 10.1097/PCC.0b013e31820aba48. PMID 21283046